CLINICAL TRIAL: NCT03668626
Title: Family-Centered Intervention for Preterm Children: Effects at School Age and Biosocial Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201801017RINA
Record Dates: First submitted 2018-08-28; First posted 2018-09-12 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Premature Birth
Keywords: intervention; effectiveness
MeSH Terms: conditions — Premature Birth | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Term infants (No Intervention): Healthy term infants
- Usual care program (UCP) (No Intervention): In-hospital and after-discharge intervention (telephone calls)
- Family-centered intervention program (FCIP) (Experimental): In-hospital and after-discharge intervention (clinic and home visits)
  Interventions: Other: Family-centered intervention program (FCIP)

INTERVENTIONS:
Other: Family-centered intervention program (FCIP) — This program included in-hospital intervention, after-discharge intervention and neonatal follow-up. Five sessions of in-hospital intervention emphasized modulation of the NICU, teaching of child developmental skills, feeding support, massage, interactional activities and parent support and education. The 7-session after-discharge intervention consisted of 4 clinic visits and 3 home visits with specific care in modulation of home environment, teaching of child developmental skills, feeding support, teaching of interactional activities, and parent support and education.
  Other Names: early intervention program
  Arms: Family-centered intervention program (FCIP)

SUMMARY:
This study is to extend our previous research to longitudinally examine the effectiveness of intervention programs (FCIP and UCP) for VLBW preterm children in Taiwan at seven years of age. Gender and maternal education level matched term children will also be included to serve as the reference group for comparison of developmental outcomes. The intervention had been delivered from birth to one year of corrected age in the previous study. Effectiveness examined will include child and parent outcomes. Primary outcome refers to measures of child neurobehavioral and neurophysiological functions. Neurobehavioral assessment includes cognitive, motor and behavioral measurement. Neurophysiological assessment refers to electroencephalogram/event-related potential examination and cognition/motor dual tasks that will be used to investigate the neurological pathways underlying the effective intervention. Secondary outcomes refer to child growth and health, and the quality of parenting measures.

DETAILED DESCRIPTION:
Preterm children present more cognitive impairments, psychological and behavioral problems, motor and coordination impairments than their term counterparts. These impairments may cause the difficulties of learning and adaptation at the school age when facing multiple and complicate environmental stimulations in preterm children. Accumulating data on early intervention for preterm infants in Eastern and Western countries have demonstrated short- to medium-term benefits on enhancing child neurodevelopment outcomes. However, rare studies have examined the effectiveness of early intervention for preterm infants and its underlying neural mechanism. To meet the contemporary concept of family centered care, we have developed a family-centered intervention program (FCIP) for preterm infants with very low birth weight (VLBW, birth weight <1,500 g) in Taiwan and have found short-term developmental benefit with respect to a usual care program (UCP) via a multi-centered, randomized controlled trial. Therefore, this three-year project is aimed to continuously follow-up the effectiveness of FCIP on child and parent outcomes in VLBW preterm infants at school age. A total of 275 VLBW preterm children (269 participants and 6 pilots) who had participated in our previous randomized controlled study and 45 term children will be assessed growth, health, neurobehavioral functions (cognition, language, motor and behaviors), electroencephalography and event-related potentials (in the resting state, cognitive inhibitory control and working memory procedures) and cognition/motor dual tasks at 7 years of age. Parents will be assessed for stress using the Parenting Stress Index/Long Form and quality of life with the World Health Organization Quality of Life- Brief Taiwan Version. The effect of early intervention for preterm children from the neonatal period to school age will provide important information to help medical professionals and public policy makers design effective intervention for Taiwanese preterm children. The continuous neurophysiological and neurobehavioral data are crucial for understanding the neurophysiological mechanisms underlying neurobehavioral changes following intervention.

ELIGIBILITY:
Inclusion Criteria:

* birth body weight < 1500 grams
* gestational age < 37 weeks
* parents of Taiwan nationality, married or together at delivery, and northern family residing in greater Taipei and southern family residing in greater Tainan, Kaohsiung, or Chiayi

Inclusion Criteria for Term infants:

* birth body weight > 2000 grams
* gestational age > 37 weeks
* parents of Taiwan nationality

Exclusion Criteria:

* severe neonatal and perinatal diseases (e.g., seizures, hydrocephalus, meningitis, grade III-IV IVH and grade II NEC)
* congenital or chromosome abnormality
* mother < 18 years, with mental retardation or history of maternal substance abuse at any time (smoking, alcohol and drug)

Terminated Criteria for Preterm infants:

* diagnosis of brain injury (e.g., PVL, stage IV ROP or greater)
* severe cardiopulmonary disease requiring invasive or non-invasive ventilator use at hospital discharge
* hospital discharge beyond 44 weeks' post-menstrual age.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Child: Neurodevelopment- The Wechsler Preschool and Primary Scale of Intelligence-Fourth Edition | 2 years
  The Wechsler Preschool and Primary Scale of Intelligence-Fourth Edition (WPPSIR-IV) measures cognitive development of children aged from 6 years to 16 years and 11 months old. The test structure of WPPSIR-IV includes 14 subscales and several levels of interpretation: verbal comprehension index, perceptual reasoning index, working memory index, processing speed index and full scale intelligence quotient. The scaled score of each subscale ranges from 1 to 19. The total scaled score is the sum of the subscale scores ranging from 10 to 190. The full scale intelligence quotient will be converted from the total scaled score with a higher value indicating a better performance.

SECONDARY OUTCOMES:
Child: Past medical history | up to 2 years
  Past 1-year medical history is recorded by parental interview.
Child: Academic performance | up to 2 years
  Parent interview
Child: Neurodevelopment - Movement Assessment Battery for Children- 2nd Edition | 2 years
  The Movement Assessment Battery for Children- 2nd Edition examines the motor performance in children aged 3 years to 16 years and 11 months. The assessment contains eight items that measure a child's performance of age-appropriate tasks in the aspects of manual dexterity, aiming and catching, and balance. The scaled score of each subscale ranges from 1 to 19. The total score is the sum of the raw scores of the subscales and can be converted to scaled score, ranging from 10 to 190, and percentile. A higher score indicates a better performance.
Child: Electroencephalogram (EEG) | 2 years
  Electroencephalogram (EEG) will be measured in the resting state for the participating children at 7 years of age.
Child: Event-related potential (ERP) | 2 years
  Event-related potential (ERP) will be measured in the cognitive inhibitory control and working memory procedures and cognition/motor dual tasks with ERP technique for the participating children at 7 years of age.
Parent function-pressure | 2 years
  Parenting Stress Index measures stress of parents of children aged 1 month to 12 years. The total score ranges from 94 to 486, with a higher score indicating a higher stress.
Parent function-quality of Life | 2 years
  World Health Organization Quality of Life- Brief Taiwan version has a total score ranging from 34 to 170. A higher score indicates a better quality of life.
Child: Behavior - Child Behavior Check List/ 4-18 | 2 years
  The Child Behavior Check List/ 4-18 is a parent-report questionnaire designed to assess the behavior problems in children at 4 to 18 years of age. The CBCL/4-18 consists of 138 items to assess child's behavioral/emotional problems. The total score ranges from 0 to 200, with a higher score indicating a worse behavior.
Child: Behavior - Swanson, Nolan, and Pelham Questionnaire, version IV | Time Frame: 1 year
  The Swanson, Nolan, and Pelham Questionnaire, version IV questionnaire examines the severity of ADHD and ODD in preschool- and school-aged children. The scale employs the direct symptom of Diagnosis and Statistical Manual of Mental Disorder-IV (DSM-IV) that consists of inattention (nine items), hyperactivity/impulsivity (nine items) of the criteria for ADHD, and the oppositional symptoms (eight items) of the criteria for ODD.
  The total score ranges from 0 to 73, a higher score indicating a worse performance.
Child: Growth - weight | up to 2 years
  weight will be assessed using an electric weight scale (kg)
Child: Growth - height | up to 2 years
  height will be assessed by the tape measure in standing position (cm)
Child: Growth - head circumference | up to 2 years
  head circumference will be assessed as the largest dimension around the head obtained with a type measure placed snugly above the ears (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Professor, Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No